CLINICAL TRIAL: NCT00001686
Title: Treatment of Children With Cancer
Brief Title: Evaluation, Treatment, and Natural History of Children and Young Adults With Cancer or Rare Diseases
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980037; 98-C-0037; NCT00445536 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Ewing's Sarcoma; Leukemia; Lymphoma; Brain Tumors; Rhabdomyosarcoma
Keywords: Leukemia; Ewing's Sarcoma; Neuroectodermal Tumors; Lymphoma, Osteosarcoma; Brain Tumors, Rhabdomyosarcoma; Lymphoma; Neoplasm; Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Leukemia; Lymphoma; Brain Neoplasms; Rhabdomyosarcoma; Neuroectodermal Tumors; Osteosarcoma; Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort A: Children and adults with cancer (or a pre-cancer syndrome or rare disease), between the age(s) of 2 years - 40 years, who present with disease manifestations of special interest to POB investigators.

SUMMARY:
This protocol is designed to evaluate children with cancer who appear to be probable candidates for future protocol entry or have disease manifestations that are of unique scientific importance or educational value.

DETAILED DESCRIPTION:
Background:

Children and adults are referred to the Pediatric Oncology Branch (POB) for possible enrollment in clinical protocols for the treatment of cancer or other rare diseases. While some children are not eligible for a specific protocol, they may present with disease manifestations that offer the potential for important new insights into the pathogenesis or clinical behavior of their underlying disease. In addition, children who have completed participation in a clinical protocol but do not currently have therapeutic protocol alternatives may continue to provide POB with important information. Diseases of interest to the POB include, but are not limited to lymphoma, brain tumors, Ewing's sarcoma, leukemia, neuroectodermal tumors, osteosarcoma, rhabdomyosarcoma, RAS-related syndromes and inherited immune disorders, amongst others. Hence, serial clinical evaluation of such patients, including the performance of clinical, laboratory, and diagnostic studies to help elucidate longitudinally the underlying disease mechanisms, and when clinically indicated standard care therapies, will assist POB meet its overall mission.

Objectives:

To be able to follow and evaluate children and adults with cancer or pre-cancer syndromes and other rare diseases referred to the Pediatric Oncology Branch who present with disease manifestations that lend themselves to clinical evaluation and are of unique scientific importance.

Eligibility:

Patients who are evaluated by the Pediatric Oncology Branch and are:

* Children and adults with cancer (or a pre-cancer syndrome or rare disease), with disease manifestations of special interest to Pediatric Oncology Branch investigators.
* Patients must be greater than or equal to 2 years and less than or equal to 40 years of age at the time of study enrollment.

Design:

The medical procedures or tests will be selected for each patient on the basis of his/her individual diagnosis (or presumed diagnosis). When clinically indicated, standard therapy will be administered and patients will be followed according to standard medical practice. Specimens may be collected for clinical care purposes only to evaluate the patient s status. No investigational tests, drugs or therapies will be administered in this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:
* A POB, CCR investigator decides that it is in the best interest of the patient and the POB, CCR for the patient to receive treatment and follow-up at the NCI/NIH.
* Children and adults with cancer (or a pre-cancer syndrome or a rare disease), between the age (s) of 2 years - 40 years (the NIH CC is not well equipped to provide optimal care to patients < 2 years of age). Note: Patients greater than or equal to 18 and less than or equal to 40 years may be evaluated on this protocol if their cancer (or precancer syndrome or rare disease) is of specific interest to the POB, CCR, NCI.
* Patients with cancer (or a pre-cancer syndrome or rare disease), who present with disease manifestations of special interest to Pediatric Oncology Branch investigators, including but not limited to, lymphoma, brain tumors, Ewing's sarcoma, leukemia, neuroectodermal tumors, osteosarcoma, rhabdomyosarcoma,RAS-related syndromes and inherited immune disorders, amongst others.
* Patient must weigh greater than or equal to 12 kg (the NIH CC is not well equipped to provide optimal care to patients < 12 kg)
* The patient, parent, guardian or their Legally Authorized Representative (LAR) is able and willing to provide informed consent.
* Patients, and when indicated, parent, guardian or LAR who are deemed sufficiently reliable to return for recommended follow-up visits.

EXCLUSION CRITERIA:

* Patients younger than 2 years of age.
* Patients weighing less than or equal to 12 kg.
* Pregnant women are excluded from enrollment onto this study because the invasive procedures and/or sedation needed to perform these may cause unnecessary harm to the unborn fetus. In the event a woman becomes pregnant while on study, she will not be removed from the study; however, no invasive clinical or research procedures will be done or cancer treatment provided during pregnancy that include unacceptable risk to the patient and/or to the unborn fetus.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adults with cancer (or a pre-cancer syndrome/rare disease), between the age(s) of 2 years - 40 years, who present with disease manifestations of special interest to POB investigators.
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 1998-03-19 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Evaluate children and adults with cancer | End of treatment
  evaluate longitudinally children and adults with cancer, pre-canceroussyndromes or rare diseases referred to the Pediatric Oncology Branch (POB) who present with disease manifestations that lend themselves to clinical evaluation and are of unique scientific importance

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1998-C-0037.html